CLINICAL TRIAL: NCT04745702
Title: Food Based Intervention Rich in Plant Components to Improve Metabolic Health in Prediabetics (FBIP) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019/00997
Record Dates: First submitted 2021-02-01; First posted 2021-02-09 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Diabetes
Keywords: Pre-diabetes; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Calorie Control Group (Other): The control group will receive for 2 calorie-restricted balanced meals per day, consisting of a portion of meat, a portion of vegetables, a portion of medium to high GI carbohydrates and prepared with refined corn oil. The control meals will be devoid of any whole legumes and will contain minimal amounts of spices. The third meal of the day and any additional snacks will be left to the free choice of the participants with calorie advice provided by study dietitian. Calorie restriction aims to reduce weight of participants by ~5%.
  Interventions: Combination Product: Low Calorie Balanced Meals
- Low-Calorie Treatment Group (Active Comparator): The treatment group will receive for 2 calorie-restricted (isocaloric with control group) meals per day containing 100 g cooked whole legumes (amounting to a total of 200 g cooked legumes, approximately 1 cup of cooked legumes)and/or certain meat analogues (textured vegetable [soy] proteins), and/or a portion of vegetables, low GI, wholegrain carbohydrates for their starch sources (rice/noodles/pasta), added spices (dried spice powder) at dietary and culinary acceptable doses and blended vegetable oil. The third meal of the day and any additional snacks will be left to the free choice of the participants with calorie advice provided by study dietitian. Calorie restriction aims to reduce weight of participants by ~5%.
  Interventions: Combination Product: Low Calorie Meals Rich in Plant Components

INTERVENTIONS:
Combination Product: Low Calorie Meals Rich in Plant Components — Twice a day reduced calorie frozen ready meals (rich in plant components) to substitute participants' two main meals/day consecutively for a period of 16 weeks.
  Arms: Low-Calorie Treatment Group
Combination Product: Low Calorie Balanced Meals — Twice a day reduced calorie frozen ready meals (balanced composition) to substitute participants' two main meals/day consecutively for a period of 16 weeks.
  Arms: Low-Calorie Control Group

SUMMARY:
The estimated prevalence of type 2 diabetes and prediabetes in Singapore will be approximately 20% and 25% respectively by the year 2035. Therefore, effective population based interventions are urgently warranted to halt this burden. Lifestyle intervention is the cornerstone of diabetes prevention and even remission. For example, dietary patterns such as the Mediterranean diet, Dietary Approaches to Stop Hypertension (DASH) diet etc. have all been shown to reduce risk of type 2 diabetes incidence. Therefore, given the successful utility of various dietary patterns, this randomized controlled trial will investigate the effectiveness of a food based dietary intervention, within an Asian dietary context, using legumes, low glycemic index (GI) starches (i.e., rice, noodles etc.), healthier vegetable oil blend as well as herbs and spices to improve various markers metabolic health, including glucose homeostasis in individuals with prediabetes.

DETAILED DESCRIPTION:
The worldwide prevalence of type 2 diabetes has increased by more than two-fold over the past three decades, with ~60% of diabetics in the world currently living in Asian countries. Type 2 diabetes occurs at a younger age and at lower body mass index (BMI < 22 kg/m2) in Asians as compared other ethnic groups. Among the various evidence based approaches to diabetes prevention, diet plays one of the most important roles. In particular, food based interventions are beginning to emerge as superior strategies in the prevention of type 2 diabetes compared to nutrient based approaches. It is important of course to align food based interventions to the cultural and region specific aspects of food choice and eating behavior if such lifestyle pattern is to be implemented in a given population. To this effect, the investigators will investigate the effects of a multiple food components in combination on metabolic health outcomes, within an Asian dietary context. This proposed study will be undertaken in prediabetics who are at greater life-time risk of developing type 2 diabetes than their normoglycemic counterparts.

Based on the current evidence, the investigators will design a food based intervention consisting of a diet rich in legumes, low GI starches (such as rice, noodles),healthier vegetable oil blends (such as rice bran, peanut, sesame seed and sunflower oils) as well as certain herbs and spices. As part of this study, each volunteer will be provided with 2 of their 3 meals per day, consisting of the above mentioned foods, for a period of 16 weeks. The control group will also be provided 2 meals per day, matched for the total calorie contents. The total calorie content of each provided meal will be approximately 500 kcal for males and 400 kcal for females. The difference in the calorie contents between the genders will be made up by using prepacked snacks. There will also be further differences in the snack types between the two intervention (treatment vs control) groups. While the treatment group will consist of healthier snacks such as seeds and wholemeal crackers, the control group snack ingredients will be made from refined flour biscuits etc. The remaining foods (free choice) during the day will be monitored regularly by the study dietitian to ensure a small calorie deficit that should lead to an approximately 5% weight loss in both intervention and control groups. Therefore, while it is expected that even the control group will achieve some metabolic health benefits during this 16 week dietary intervention (indirectly due to weight loss), the investigators anticipate that the treatment group will attain greater benefits as compared to the control group, due to the differences in their food constituents. The effects of dietary interventions on metabolic health will be assessed at every 4-8 week intervals. The primary outcome measures will include several markers of glucose homeostasis (including HbA1c, fasting glucose, fasting insulin and a 2-hr oral glucose tolerance test [OGTT]). The secondary outcomes will include blood lipid profile, fructosamine, adiponectin, markers of oxidative stress and chronic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Male or Female• Age between 45-75 years
* Body mass index 19.5-32.0 kg/m2
* Deemed to be prediabetic based on meeting any 1 of 3 following criteria:1. Fasting blood glucose >5.5 mmol/l and <7.0 mmol/l2. Oral glucose tolerance test (OGTT) level >/=7.8 mmol/l and </=11.0 mmol/l3. Haemoglobin A1c (HbA1c) level >/=5.7 and </=6.4%.

Exclusion criteria:

* Smoking
* Having allergies or intolerances to any common food ingredients including eggs, fish, milk, peanuts, and tree nuts, shellfish, soya, wheat, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, natural food colourings or flavourings, etc.
* Following special diets or having intentional dietary restrictions (e.g, vegetarians/vegans)
* Not willing to adhere to diet modification as in the study protocol
* Not willing to stop any strenuous activity during or within 24 hours of test days (for those actively participating in sports at the competitive and/or endurance levels)
* Having glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Having alcohol consumption on > 4 days per week with ≥ 6 alcoholic drinks per week
* Having sustained elevation of blood pressure (>160/95 mm Hg)
* Having previously undergone any gastrointestinal surgery or having history of gastrointestinal disorders
* Having a history of heart, liver, kidney, blood disorders (e.g., thalassemia) or thyroid dysfunctions
* Diabetic
* Having history of tuberculosis, HIV, Hepatitis B or Hepatitis C infections
* Having any prescription medication or any other alternative medicines or supplements which may interfere with study measurements in the in the opinion of the study investigators
* Having antibiotics or suffering from diarrhea within the last 3 months
* Having donated blood within 4 weeks of study participation
* Having poor veins or having history of severe vasovagal syncope (blackouts or fainting) from blood draws
* Having more than 5% weight loss or gain over the past 3 months
* For female volunteers: menstruation within past 12 months or being on hormone replacement therapy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-08-09 (Estimated); Study Completion 2022-08-09 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 16 weeks
  mmol/mol (%)
Fasting glucose | 16 weeks
  mmol/L
Fasting insulin | 16 weeks
  pmol/L
Oral Glucose Tolerance Test | 16 weeks
  mmol/L

SECONDARY OUTCOMES:
Blood Lipid Profile (HDL, LDL, Total Cholesterol, Triglyceride) | 16 weeks (from first to final measurement visits), measured every 4 weeks
  mmol/L
Fructosamine | 16 weeks (from first to final measurement visits), measured every 4 weeks
  µmol/L
Plasma Adiponectin | 16 weeks (from first to final measurement visits), measured every 4 weeks
  μg/mL
Oxidised LDL | 16 weeks (from first to final measurement visits), measured every 4 weeks
  ng/mL
C-Reactive Protein | 16 weeks (from first to final measurement visits), measured every 8 weeks
  mg/L
IL-6 (interleukin 6) | 16 weeks (from first to final measurement visits), measured every 8 weeks
  pg/mL
TNF (Tumor Necrosis Factor - alpha) | 16 weeks (from first to final measurement visits), measured every 8 weeks
  pg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu X, Tjahyo AS, Volchanskaya VSB, Wong LH, Lai X, Yong YN, Osman F, Tay SL, Govindharajulu P, Ponnalagu S, Tso R, Teo HS, Khoo K, Fan H, Goh CC, Yap CPL, Leow MK, Henry CJ, Haldar S, Lim KJ. A legume-enriched diet improves metabolic health in prediabetes mediated through gut microbiome: a randomized controlled trial. Nat Commun. 2025 Jan 22;16(1):942. doi: 10.1038/s41467-025-56084-6. PMID 39843443